## Evaluation of Efficacy of LANAP and Adjunctive LLLT Application in the Treatment of Periodontitis: A Randomized Controlled Clinical Study

The statistical analysis of the data obtained in the study was performed using statistical package program (SPSS version 22). While clinical, laboratory and radiographic data were presented and evaluated, descriptive statistical terms such as arithmetic mean, standard deviation (ss), median, minimum (min) and maximum (max) values were used. In order to determine the statistical distribution of clinical periodontal parameters, biochemical and radiographic data, Kolmogorov-Smirnov and Shapiro-Wilk tests were performed. In the study, while repeated measures ANOVA was applied in the intra-group comparison of dependent variables that were normally distributed, one-way ANOVA was applied in the comparison between the groups. If the dependent variables were not normally distributed, the Friedman test was used for intragroup comparison, followed by the Wilcoxon test for multiple comparisons. Kruskal-Wallis test was used for intergroup comparison, followed by Dunn test for multiple comparisons. The statistical significance of the results was evaluated as p <0.05.